CLINICAL TRIAL: NCT04151212
Title: A Phase I Clinical Trial for BAT5906(Single-dose;for Injection) on Safety and Pharmacokinetics for Patients With Age-related Macular Degeneration
Brief Title: A Phase I Clinical Trial of BAT5906 Injection in Patients With Wet Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAT5906-001-CR
Record Dates: First submitted 2019-11-04; First posted 2019-11-05 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2019-10

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAT5906 injection (Experimental): Single dose escalation starting from 0.3mg. Route of administration: intravitreal injection.
  Interventions: Drug: BAT5906 injection

INTERVENTIONS:
Drug: BAT5906 injection — Signal dose escalation starting from 0.3mg. Route of administration: intravitreal injection
  Other Names: No Other Intervention Names

SUMMARY:
A Phase I Clinical Trial for BAT5906(single-dose;for injection) on Safety and Pharmacokinetics for Patients with Age-related macular degeneration.

DETAILED DESCRIPTION:
The primary objective: To evaluate the safety and Pharmacokinetics of BAT5906 (single-dose Ophthalmic Intracireal Iinjection) in patients wAMD , when the injection dosage escalates.

The Secondary objective: To evaluate the immunogenicity profile of BAT5906; To evaluate the pharmacodynamics and therapeutic efficacy profile of BAT5906.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 50-80 years old .
* Signing the informed consent form and able and willing to comply with all treatment and follow-up study procedures.
* The study eye must meet all the following inclusion criteria: To be diagnosed as wet age related macular degeneration, and there are still active lesions currently;Total lesion size of ≤30mm2( 12 disc areas);Best corrected visual acuity ≤70 Early Treatment of Diabetic Retinopathy ;Study letters (≤20/40) in the study eye.
* Best corrected visual acuity ≥34 Early Treatment of Diabetic Retinopathy Study letters (≥20/200) . in the non-study eye.

Exclusion Criteria:

* There are atrophy of the ground pattern involving the fovea, scar or fibrosis, macular anterior membrane, rigid exudation under dense fovea, RPE tear in the study eye.
* Retinal hemorrhage ≥4 disc area in the study eye.
* Dioptric media turbid or the pupil cannot be dilated were significant interference with the detection of vision, the evaluation of the anterior segment and fundus in the study eye.
* Evidence of ocular disease other than exudative AMD in the study eye that may confound the outcome of the study (e.g.,Retinal vein occlusion, uveitis, vascular striatum, pathological myopia, retinal detachment, macular hole, toxoplasmosis, optic nerve disease etc).
* History of vitrectomy surgery\macular transposition\glaucoma filtration in the study eye.
* Photodynamic therapy(PDT), in macular area laser photocoagulation therapy, transpermary hyperthermia(TTT), and other operations for AMD within 3 months prior to screening visit in the study eye.
* History of extraocula surgeryr within 1 months or cataract surgery within 3 months prior to screening visit in the study eye.
* Aphakia(exclusive of intraocular lens) or rupture of posterior capsule( within1 months prior to the YAG laser retrovesiculotomy (after the artificial crystal), was excluded) in the study eye.
* APD in the study eye or pseudocyst stripping syndrome in either eye.
* Intravitrea or Systemicl anti-VEGF injection (ranibizumab, aflibercept, bevacizumab or Conbercept etc) in either eye within 3 months prior to screening visit.
* Under the conjunctiva,intravitreal or periocular corticosteroid, within 3 months prior to screening visit in either eye.
* vitreous hemorrhage within 3 months prior to screening Visit in either eye.
* Ocular or periocular infection in either eye.
* History of glaucoma in either eye.
* Visudyne (verteporfin) photodynamic therapy within 1 months prior to screening Visit in non-study eye.
* Currently in use or may be required to use systemic drugs that cause crystal toxicity or retinal toxicity, such as Deferoxamine, chloroquine/ hydroxychloroquine, phenothiazine and ethambutol or tamoxifen etc.
* Have an allergic reaction or history of allergic reactions to fluorescein sodium and indocyanine green, an allergic history to therapeutic or diagnostic protein products, an allergic reaction to more than two drugs or non-drug factors, or allergic reactions to any monoclonal antibody.
* Patients with diabetic retinopathy or the diabetic patient who have glycosylated? hemoglobin>10%.
* Patients who have undergone any surgical operation within 1 month prior screening; or/and there are unhealed wounds, ulcers, fractures etc.
* Systemic infectious diseases with clinical significance requiring oral, intramuscular or Patients withintravenous administration.
* Myocardial infarction, cerebral infarction and angina pectoris within 6 months prior to screening visit.
* Patients with active disseminated intravascular coagulation and obvious bleeding tendency were screened within 3 months before the screening, or they were treated with anticoagulant and antiplatelet therapy other than aspirin/NSAIDs within 14 days before the screening.
* Patients with Systemic immune disease ,including but not limited to:

hyperthyroidism, hypothyroidism,vitiligo, dry-syndrome, ankylosing spondylitis, systemic nephritis, human immunodeficiency virus (HIV).

* Blood pressure control is not ideal or pre-hypertension.
* Any uncontrollable clinical problems (Serious mental, nervous, cardiovascular and respiratory diseases and malignant tumors).
* Abnormal liver and kidney function.
* Blood coagulation is abnormal.
* Patients with AIDS, syphilis or active hepatitis.
* Women are not using effective contraception or in pregnancy,lactation.
* Clinical trials of any trial medication or any other experimental or experimental therapy may be performed within 3 months prior to screening.
* Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 2 weeks
  Safety and tolerability endpoint
Maximum tolerated dosed(MTD) | 0-70days
  Safety and tolerability endpoint
Area under the curve(AUC0-t, AUC0-inf) | 0-70days
  Pharmacokinetic endpoint Pharmacokinetic endpoint
Maximum serum drug concentration(Cmax) | 0-70days
  Pharmacokinetic endpoint Pharmacokinetic endpoint
Half-life period(t1/2) | 0-70days
  Pharmacokinetic endpoint
Maximum serum drug time(Tmax) | 0-70days
  Pharmacokinetic endpoint
Plasma clearance(CL) | 0-70days
  Pharmacokinetic endpoint

SECONDARY OUTCOMES:
Anti-drug antibodies(ADA) | 0-70days
  Immunogenic endpoint
Best correct vision(BCVA) | 0-70days
  Effective endpoint
Central Retinal thickness(CRT) | 0-70days
  Effective endpoint
VEGF concentration | 0-70days
  Pharmacodynamics endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, China